CLINICAL TRIAL: NCT05802264
Title: A 3-part Study of ABCI: a Randomized, Double-blind, Placebo-controlled, Single-ascending Dose Phase 1a Study in Healthy Volunteers (Part A), a Randomized, Double-blind, Placebo-controlled, 14- and 28-day Multiple-ascending Dose Phase 1a Study in Healthy Volunteers (Part B), and a 28-day Open-Label Phase 1b Study in Subjects with Cystic Fibrosis (Part C)
Brief Title: Study to Assess Amphotericin B Cystetic for Inhalation (ABCI) Doses in Healthy Volunteers & People with Cystic Fibrosis
Acronym: ABCI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cystetic Medicines, Inc. (Industry)
Collaborators: DevPro Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM001001
Record Dates: First submitted 2023-02-28; First posted 2023-04-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part A Healthy Volunteer (Experimental): Subjects will be assigned to one of six planned dose cohorts and receive single doses of ABCI (0.5mg, 1.0mg, 2.0mg, 4.0mg, 6.0mg, 10.0mg). In each cohort, six subjects will receive ABCI and 2 will receive placebo
  Interventions: Combination Product: ABCI; Combination Product: Placebo
- Part B Healthy Volunteer (Experimental): Subjects will be assigned to one of three planned dose cohorts and receive a loading dose and multiple ascending doses of ABCI (loading dose 1.5mg/0.5mg daily, loading dose 6.0mg/2.0 daily, loading dose 10.0mg/4.0mg daily). In each cohort, six subjects will receive ABCI and 2 will receive placebo.
  Interventions: Combination Product: ABCI; Combination Product: Placebo
- Part C People with Cystic Fibrosis (Experimental): Subjects will be assigned to one of two planned dose cohorts of ABCI (loading dose 1.5 mg/0.5 mg daily, loading dose 6.0mg/2.0mg daily, loading dose 10.0mg/4.0mg daily) for a total of 28 days of open-label study drug administration. Up to 36subjects with CF, including 2 sentinels subjects not on cystic fibrosis transmembrane conductance regulator (CFTR) modulators will be enrolled. The 2 sentinel subjects will receive the medium dose/regimen. If the medium dose/regimen is tolerated, the remaining subjects with CF may receive the low, medium, high dose/regimen of ABCI and may be either on CFTR modulators or not on CFTR modulators. It is anticipated that approximately 24 subjects will be enrolled as follows: 8 high, 8 medium, and 8 low dose/regimen.
  Interventions: Combination Product: ABCI

INTERVENTIONS:
Combination Product: ABCI — Subjects will receive ABCI via oral inhalation
  Other Names: Amphotericin B Cystetic for Inhalation
Combination Product: Placebo — Subjects will receive ABCI via oral inhalation
  Arms: Part A Healthy Volunteer; Part B Healthy Volunteer

SUMMARY:
This is a 3-part, single-ascending dose Phase 1a randomized, double-blind, placebo-controlled study in healthy volunteers (Part A) and multiple-ascending dose Phase 1a randomized, double-blind, placebo-controlled study in healthy volunteers (Part B), and a Phase 1b open-label study in subjects with CF (Part C) to assess the safety, tolerability, PK, and preliminary efficacy of ABCI. Subjects will be evaluated for eligibility during Screening within 30 days prior to Day 1 (Randomization; Visit 3). In Parts A and B, eligible healthy volunteers may be enrolled in the study and randomly allocated to treatment with ABCI or placebo as described below. In Part C, eligible subjects with CF may be enrolled in the study and receive treatment with ABCI as described below. Approximately 72 healthy subjects total will be randomized to 9 cohorts (48 subjects in 6 cohorts in Part A, 24 subjects in 3 cohorts in Part B) and approximately 36 subjects with CF will receive the low dose, medium dose (2 sentinel subjects), or high dose of ABCI in Part C.

ELIGIBILITY:
Inclusion Criteria:

Part A and Part B: Each subject must meet the following criteria to be enrolled in Part A and Part B of this study.

* Subject has signed, dated, and received a copy of the IRB/IEC-approved written ICF.
* Subject is male or female aged ≥18 to ≤55 years.
* Subject has a BMI between 18 and 32 kg/m2
* Subject has an FEV1 of >90% of predicted normal value
* Subject has normal or clinically acceptable physical examination, vital signs, clinical laboratory values, and ECG at Screening.
* Female subjects must be of non-childbearing potential or male/female subjects of childbearing potential agree to use highly effective contraception/preventive exposure measures

Part C: Each subject must meet the following criteria to be enrolled in Part C of this study.

* Subject has signed, dated, and received a copy of the IRB/IEC-approved written ICF.
* Age 16 years or older
* Confirmed diagnosis of CF, including sweat chloride >60 mM.
* Subject is either: Being treated with an approved CFTR modulator for at least 28 days prior to Screening, or Not being treated with a CFTR modulator
* FEV1:
* For subjects on CFTR modulators: FEV1 ≥40% and ≤90%
* For subjects not on CFTR modulators: FEV1 ≥40% and ≤100%
* Stable CF disease and treatment regiment
* Female subjects must be of non-childbearing potential or male/female subjects of childbearing potential agree to use highly effective contraception/preventive exposure measures

Exclusion Criteria:

Part A and Part B: Any subject who meets any of these criteria must be excluded from Part A and Part B of this study:

* Subject has history or evidence of any clinically significant pulmonary condition
* Subject has history or evidence of any clinically significant diseases or conditions
* Subject has history of malignancy of any type
* Subject has an active COVID-19 infection within 4 weeks
* Subject is positive for human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C antibodies, or has a positive QuantiFERON®-tuberculosis Gold (QFT-G) test for tuberculosis at Screening
* Subject has a self-reported lower respiratory tract infection within 6 weeks
* Subject has evidence of any active or suspected bacterial, viral, fungal or parasitic infections within the past 4 weeks
* A subject who is an active smoker or a former smoker
* Subject has history of alcohol or drug abuse in the past year
* Subject has tested positive for drugs (including cannabis), nicotine/cotinine, and/or alcohol use at Screening, subject has consumed alcohol within 24 hours prior to Visit 3
* Subject has participated in any clinical study or had been treated with any investigational drugs within 28 days or 5 half-lives
* Female subject who is pregnant or breastfeeding.
* Subject has any episode of paradoxical bronchospasm in the past 12 months.
* Subject has pacemaker; is not in sinus rhythm; has a corrected QT interval (QTc; using Fridericia's [QTcF] formula) of >450 ms (for males) and >470 ms (for females); or has a left bundle branch block or bifascicular block.
* Subject has a pulse <40 or >100 bpm; systolic blood pressure >140 mmHg, or diastolic blood pressure >90 mmHg at Screening
* Subject has Type I or II diabetes requiring medication.
* Subject has received any vaccine within 30 days prior to Day 1.
* Subject has received any of the following immunosuppressant therapies within 6 months prior to Screening: imatinib, ambrisentan, azathioprine, cyclophosphamide, cyclosporine A, bosentan, or methotrexate.
* Subject has received any antibody or therapeutic biologic product during the 6 months prior to Screening.
* Subject has received any oral, intravenous, or intramuscular steroid within 4 weeks prior to Screening. Intrathecal or intraarticular steroids are permitted.
* A subject who is not vaccinated with the COVID-19 vaccine with appropriate window from last dose of vaccine to Screening per local guidelines, policies, and availability within 30 days prior to Day 1.

Part C: Any subject who meets any of these criteria must be excluded from Part C of this study:

* History of any illness or any clinical condition that might confound the results of the study or pose an additional risk in administering study drug(s) to the subject.
* Any of the following abnormal laboratory tests: Hemoglobin, Total bilirubin, liver enzymes or creatine clearance
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy for sinopulmonary disease within 28 days before the screening visit.
* An acute illness not related to CF within 14 days before the first dose of study drug.
* Subject has an active COVID-19 infection within 4 weeks prior to screening.
* Ongoing or prior participation in a study of an investigational treatment within 28 days or 5 terminal half-lives (whichever is longer) before screening.
* Female subject who is pregnant or breastfeeding.

Please refer to study protocol for the complete inclusion/exclusion criteria list.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs), and Serious Adverse Events (SAEs) | up to 10 weeks
  The safety and tolerability of ABCI following oral inhalation of single and multiple ascending doses in healthy subjects (Parts A and B), and in people with Cystic Fibrosis (Part C) will be assessed

SECONDARY OUTCOMES:
Pharmacokinetics (PK) Profile - SAD Cmax | 1 day
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: Observed maximum concentration (Cmax)
Pharmacokinetics (PK) Profile - SAD Tmax | 1 day
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: time to reach maximum concentration (Tmax)
Pharmacokinetics (PK) Profile - SAD AUC0-24 | 1 day
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: Area under the concentration-time curve from time 0 to 24 hours post-dose (AUC0-24)
Pharmacokinetics (PK) Profile - SAD AUClast | 1 day
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast)
Pharmacokinetics (PK) Profile - SAD AUCinf | 1 day
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: Area under the concentration-time curve from the time of dosing extrapolated to infinity (AUCinf)
Pharmacokinetics (PK) Profile - SAD AUCtau | Up to 28 days
  Pharmacokinetics Characteristics in Single Ascending Dose HV Subjects: Area under the concentration- concentration-time curve over the dosing interval (AUCtau)
Pharmacokinetics (PK) Profile - MAD Cmax | Up to 28 days
  Pharmacokinetics Characteristics in Multiple Ascending Dose HV Subjects: Observed maximum concentration (Cmax)
Pharmacokinetics (PK) Profile - MAD Tmax | Up to 28 days
  Pharmacokinetics Characteristics in Multiple Ascending Dose HV Subjects: time to reach maximum concentration (Tmax)
Pharmacokinetics (PK) Profile - MAD AUC0-24 | Up to 28 days
  Pharmacokinetics Characteristics in Multiple Ascending Dose HV Subjects: Area under the concentration-time curve from time 0 to 24 hours post-dose (AUC0-24)
Pharmacokinetics (PK) Profile - MAD Plasma AmB assessments | Up to 84 days
  Pharmacokinetics Characteristics in Multiple Ascending Dose HV Subjects: Plasma AmB assessments
Pharmacokinetics (PK) Profile - MAD AmB concentrations in BAL fluid | Up to 29 days
  Pharmacokinetics Characteristics in Multiple Ascending Dose HV Subjects: AmB concentrations in BAL fluid after study drug administration
AmB concentrations - Subjects with CF | Through 42 days
  Cumulative effect on pre-dose AmB concentrations through Day 29 and assessment of washout through Day 42

OTHER OUTCOMES:
ppFEV1 - Subjects with CF | Up to 42 days
  Absolute change in percent-predicted morning pre-dose forced expiratory volume in 1 second (ppFEV1) from baseline to Day 29 and from Day 29 to Day 42
LCI - Subjects with CF | Up to 42 days
  Absolute change in Lung Clearance Index (LCI) (where available)
Questionnaire - Subjects with CF | Up to 42 days
  Absolute change in Cystic Fibrosis Questionnaire Revised (CFQ-R) in Subjects with Cystic Fibrosis: Revised (CFQ-R) respiratory domain score from baseline to Day 29 and to Day 42 where scores range from 0 to 100, with higher scores indicating better health.
ppFVC - Subjects with CF | Up to 42 days
  Absolute change in percent-predicted morning pre-dose forced vital capacity (ppFVC) from baseline to Day 29 and from Day 29 to Day 42
FVC - Subjects with CF | Up to 42 days
  Absolute change in morning pre-dose FVC from baseline to Day 29 and from Day 29 to Day 42 (mLs)
FEV1 - Subjects with CF | Up to 42 days
  Absolute change in morning pre-dose FEV1 from baseline to Day 29 and from Day 29 to Day 42 (mLs)
DLCO - Subjects with CF | Up to 29 days
  Absolute change in diffusing capacity of the lungs for carbon monoxide (DLCO [expressed as percent-predicted corrected for hemoglobin]) from baseline to Day 29
Body weight - Subjects with CF | Up to 42 days
  Absolute change in body weight from baseline to Day 29 and from Day 29 to Day 42
% solids in sputum - Subjects with CF | Day 29
  Absolute change in % solids in sputum from baseline (optional)
FRI biomarkers - Subjects with CF | Up to 28 days
  Change from baseline in Functional Respiratory Imaging (FRI) biomarkers, including but not limited to airway wall volume, mucus plug volume, and blood vessel volume (where available)
IVIVC - chloride secretion - Subjects with CF | Up to 42 days
  Change in chloride secretion in response to AmB in vitro in primary cultured nasal epithelial cells
IVIVC - FEV1 - Subjects with CF | Up to 42 days
  Comparison of change from baseline FEV1 (ppFEV1 and absolute FEV1) (Day 29) and change in chloride secretion in response to AmB in vitro in primary cultured nasal epithelial cells
IVIVC - ASL pH - Subjects with CF | Up to 42 days
  Change in ASL pH in response to AmB in vitro in primary cultured nasal epithelial cells
IVIVC - FEV1 & ASL pH - Subjects with CF | Up to 29 days
  Comparison of change from baseline FEV1 (ppFEV1 and absolute FEV1) (Day 29) and ASL pH in response to AmB in vitro in primary cultured nasal epithelial cells

CONTACTS AND LOCATIONS:
Overall Officials: Martin Burke, MD, PhD, Study Chair — Founder of cystetic Medicines
Locations (5):
- Australia (4):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Westmead Hospital, Westmead, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Monash Medical Centre, Clayton, Victoria
- New Zealand Clinical Research, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No